CLINICAL TRIAL: NCT06037746
Title: Immediate Effects of Myofascial Release Techniques on Balance in Young Adults With Pes Planus: A Single Blind, Randomized Controlled Pilot Study
Brief Title: Immediate Effects of Myofascial Release Techniques on Balance in Young Adults With Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PP001
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Flat Foot
Keywords: Pes Planus; Myofascial Release; Postural Balance; Randomized Controlled Trial
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Graston Group (Experimental): Miyofascial release was performed by graston tool on the entire plantar fascia.
  Interventions: Other: Graston
- Percussive Massage Group (Experimental): Miyofascial release was performed by theragun tool on the entire plantar fascia.
  Interventions: Other: Percussive massage
- Control Group (No Intervention): No application has been made.

INTERVENTIONS:
Other: Graston — For the application, the individual was asked to lie face down, flex the knee to 90 degrees and release the ankle. The therapist took a position next to the individual on the side to be treated. Application was applied to the entire plantar fascia for 10 minutes in the longitudinal, vertical and oblique directions.
  Arms: Graston Group
Other: Percussive massage — For the application, the individual was asked to lie face down, flex the knee to 90 degrees and release the ankle. The therapist took a position next to the individual on the side to be treated. Application was applied to the entire plantar fascia for 5 minutes in all directions without being bound to a single direction.
  Arms: Percussive Massage Group

SUMMARY:
The plantar fascia is a thick, multi-layered, non-elastic fibrous tissue band that extends along the plantar surface of the foot.The configuration of the plantar fascia is generally considered as a dense, longitudinally arranged fiber band divided into medial, central, and lateral components. The most significant functional role of the plantar fascia is to maintain the arch structure of the foot, providing a stable support base while standing and absorbing dynamic reaction forces during walking.Pes planus is a rather general term with many definitions. Staheli described pes planus as a "foot with a broad base of support," commonly known as flatfoot in layman's terms. In a study involving 80 female participants aged 65 and older, 90% of foot deformities observed while standing were identified as pes planus. Generally, pes planus is a condition characterized by excessive pronation of the rear part of the foot and a lowering of the medial longitudinal arch. During the push-off phase of walking, the pronation moment generated by the ground reaction force flattens the arch as the subtalar joint rotation combines. The shift in position in the talus bone causes the navicular bone to drop. The plantar calcaneonavicular ligament tightens, and the tibialis posterior muscle lengthens. Abnormalities in the bones of the foot, dysfunction of the tibialis posterior muscle, Achilles tendon shortening, or muscle weakness can contribute to pes planus. Individuals with pes planus may experience foot and leg pain with exercise, physical activity, and prolonged walking, which can limit their level of physical activity. Research has examined the relationship between pes planus and various physical parameters, and it has been found that one of these parameters, balance, is negatively affected by the presence of pes planus.

DETAILED DESCRIPTION:
Participant information, including age, gender, height, body weight, and body mass index, was recorded using a general form. Dynamic and static balance was assessed before and after the interventions in the study groups. Three specialist physiotherapists conducted measurements and evaluations (navicular drop, static and dynamic balance). The assessing physiotherapist remained consistent throughout, and they were unaware of the participant groups. An expert in manual therapy administered the MRTs. Statistical analysis was performed by a separate researcher uninvolved in the practical aspects of the study.

ELIGIBILITY:
Inclusion Criteria:

* volunteering for study participation,
* being between the ages of 18-25
* presence of pes planus.

Exclusion Criteria:

* Presence of orthopedic conditions other than pes planus,
* having a history of lower extremity surgery
* presence of neurological or rheumatological disorders,
* having a problem with vision or hearing
* participating in regular physical activity (>150 min/week)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Static Balance Test | Baseline and after immediately after intervention
  The static balance level of individuals was measured with the Flamingo Balance Test, a valid and reliable instrument. It was recorded how many times the individual fell or broke the test while trying to balance on one leg for 1 minute on a 15 cm long, 4 cm wide wooden plate. During this period, each time the test was stopped, the timer was also stopped, and the timer was restarted after the individual repositioned. The test was repeated 3 times, and the average value was recorded.
Dynamic Balance Test | Baseline and after immediately after intervention
  The dynamic balance level of individuals was measured with the "Y" Balance Test, a valid and reliable instrument, and their dominant extremities were evaluated. While trying to balance on one foot at the midpoint of the assembly, the individual was asked to reach forward with the other foot in the anterior, posteromedial, and posterolateral directions and touch the tip of the toe. The test was repeated 3 times in each direction, and the average value was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Gelisim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.